CLINICAL TRIAL: NCT00374764
Title: Randomized Double Blind Comparison of Applied Behavioral Analysis Versus ABA and Risperidone
Brief Title: Comparison of Applied Behavioral Analysis (ABA) Versus ABA and Risperidone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IND #58033
Record Dates: First submitted 2006-09-07; First posted 2006-09-11 (Estimated); Last update posted 2007-02-16 (Estimated); Status verified 2002-06

CONDITIONS: Autistic Disorder
Keywords: Autism, Applied Behavioral Analysis, Risperidone
MeSH Terms: conditions — Autistic Disorder | interventions — Risperidone

INTERVENTIONS:
Drug: Risperidone
Behavioral: ABA

SUMMARY:
Hypotheses:

1. Preschool children with autism spectrum disorders (ASDs) who undergo ABA treatment only will demonstrate significantly better outcomes compared to an age and severity matched control group without ABA treatment.
2. Preschool children with ASDs who undergo ABA in combination with risperidone will demonstrate significantly better outcomes compared to age and severity matched children who are receiving ABA alone.
3. Young age, cognitive development and attentional abilities at baseline will be predictive of good socio-emotional and neuropsychological outcomes after ABA treatment.
4. At baseline, children with ASDs will show significantly lower performances on measures of cognitive, neuropsychological, and socio-emotional functioning than age-matched typically developing controls.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of autism or severe pervasive developmental disorder (PDD) not otherwise specified (NOS) according to the Autism Diagnosis Interview-Revised (ADI-R)
* Aged 2.6 to 5.0.

Exclusion Criteria:

* Fragile X or metabolic etiology of PDD symptoms
* Diagnosis of other central nervous system (CNS) disorders
* Chronic serious medical problems

Ages: 30 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60
Dates: Start 2000-07; Study Completion 2002-06

CONTACTS AND LOCATIONS:
Overall Officials: Joan Luby, MD, Principal Investigator — Washington University Medical School
Locations (1):
- Early Emotional Development Program, St Louis, Missouri, United States

REFERENCES:
- [Background] Bachevalier, J. (1991). Memory loss and socio-emotional disturbances following neonatal damage of the limbic system in monkeys: An animal model for childhood autism. In C. Tamminga & S. Schulz (Eds.). Advances in Psychiatry and Psychopharmacology (pp. 129-140). New York: Raven Press.
- [Background] Baron-Cohen S, Cox A, Baird G, Swettenham J, Nightingale N, Morgan K, Drew A, Charman T. Psychological markers in the detection of autism in infancy in a large population. Br J Psychiatry. 1996 Feb;168(2):158-63. doi: 10.1192/bjp.168.2.158. PMID 8837904
- [Background] Bauman, M. & Kemper, T.L. (1988). Limbic and cerebellar abnormalities: Consistent findings in infantile autism. Journal of Neuropathology and Experimental Neurology, 47, 369.
- [Background] Black JE. How a child builds its brain: some lessons from animal studies of neural plasticity. Prev Med. 1998 Mar-Apr;27(2):168-71. doi: 10.1006/pmed.1998.0271. PMID 9578989
- [Background] Butterworth, G. & Jarrett, N. (1991). What minds have in common is space: Spatial mechanisms serving joint visual attention in infancy. British Journal of Developmental Psychology, 9. 55-72.
- [Background] Charman T, Swettenham J, Baron-Cohen S, Cox A, Baird G, Drew A. Infants with autism: an investigation of empathy, pretend play, joint attention, and imitation. Dev Psychol. 1997 Sep;33(5):781-9. doi: 10.1037//0012-1649.33.5.781. PMID 9300211
- [Background] Chugani HT. A critical period of brain development: studies of cerebral glucose utilization with PET. Prev Med. 1998 Mar-Apr;27(2):184-8. doi: 10.1006/pmed.1998.0274. PMID 9578992
- [Background] Chugani HT, Phelps ME. Maturational changes in cerebral function in infants determined by 18FDG positron emission tomography. Science. 1986 Feb 21;231(4740):840-3. doi: 10.1126/science.3945811.
- [Background] Courchesne E, Press GA, Yeung-Courchesne R. Parietal lobe abnormalities detected with MR in patients with infantile autism. AJR Am J Roentgenol. 1993 Feb;160(2):387-93. doi: 10.2214/ajr.160.2.8424359.
- [Background] Damasio AR, Maurer RG. A neurological model for childhood autism. Arch Neurol. 1978 Dec;35(12):777-86. doi: 10.1001/archneur.1978.00500360001001. PMID 718482
- [Background] Dawson G, Adams A. Imitation and social responsiveness in autistic children. J Abnorm Child Psychol. 1984 Jun;12(2):209-25. doi: 10.1007/BF00910664. PMID 6725782
- [Background] Dawson, G. & Castelloe, P. (1995). Autism. In C.E. Walker & M.C. Roberts (Eds.). Handbook of Clinical Child Psychology. New York. Plenum Press.
- [Background] Dawson G, Klinger LG, Panagiotides H, Lewy A, Castelloe P. Subgroups of autistic children based on social behavior display distinct patterns of brain activity. J Abnorm Child Psychol. 1995 Oct;23(5):569-83. doi: 10.1007/BF01447662. PMID 8568080
- [Background] Dawson, G. & Lewy, A. (1989). Reciprocal subcortical-cortical influences in autism: The role of attentional mechanisms. In G. Dawons (Ed.), Autism: Nature, Diagnosis, and Treatment (pp. 144-173). New York: Guilford Press.
- [Background] Dawson G, Meltzoff AN, Osterling J, Rinaldi J. Neuropsychological correlates of early symptoms of autism. Child Dev. 1998 Oct;69(5):1276-85. PMID 9839415
- [Background] Dawson, G., Warrenburg, S. & Fuller, P. (1996. Early intervention in autism. In M.J. Guralnick (Ed.), The Effectiveness of Early Intervention. Baltimore, MD: Paul Brookes Publishing Co.
- [Background] Dawson G, Warrenburg S, Fuller P. Cerebral lateralization in individuals diagnosed as autistic in early childhood. Brain Lang. 1982 Mar;15(2):353-68. doi: 10.1016/0093-934x(82)90065-7. No abstract available. PMID 7074350
- [Background] Diamond, A. & Goldman-Rakic, P.S. (1985). Evidence for involvement of prefrontal cortex in cognitive changes during the first year of life: comparison of human infants to rhesus monkeys on a detour task with transparent barrier. Society for Neurosciences Abstracts (Part II), 11, 832.
- [Background] Diamond, A. & Goldman-Rakic, P.S. (1986). Comparative development in human infants and infant rhesus monkeys on cognitive functions that depend on the prefrontal cortex. Society of Neurosciences Abstracts, 12, 742.
- [Background] Fenske, E.D., Zalenski, S., Krantz, P.J., & McClannahan, L.E. (1985). Age at intervention and treatment outcome for autistic children in a comprehensive intervention program. Analysis and Intervention in Developmental Disabilities, 5, 49-58.
- [Background] George MS, Costa DC, Kouris K, Ring HA, Ell PJ. Cerebral blood flow abnormalities in adults with infantile autism. J Nerv Ment Dis. 1992 Jul;180(7):413-7. doi: 10.1097/00005053-199207000-00002. PMID 1624921
- [Background] Gilliam, J.E. (1995). Gilliam Autism Rating Scale, Austin, TX: PRO-ED, Inc.
- [Background] Goldman-Rakic, P.S. (1987). Circuitry of primate prefrontal cortex and regulation of behavior by representational knowledge. In F. Plum & V. Mountcastle (Eds.), Handbook of Physiology, 5, 373-417.
- [Background] Goldsmith, H.H. & Rothbart, M.K. (1996). The Laboratory Temperament Assessment Battery, Locomotor Version 3.0. Madison, Wisconsin: Department of psychology, University of Wisconsin.
- [Background] Pine E, Luby J, Abbacchi A, Constantino JN. Quantitative assessment of autistic symptomatology in preschoolers. Autism. 2006 Jul;10(4):344-52. doi: 10.1177/1362361306064434. PMID 16908478